CLINICAL TRIAL: NCT04537078
Title: Progestin Primed Double Stimulation Protocol Versus Flexible GnRH Antagonist Protocol in Poor Responders
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: El Shatby University Hospital for Obstetrics and Gynecology (Other)
Responsible Party: Principal Investigator, Aly Hussein, Assistant lecturer, University of Alexandria, El Shatby University Hospital for Obstetrics and Gynecology
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0201350
Record Dates: First submitted 2020-08-28; First posted 2020-09-03 (Actual); Results first posted 2022-02-17 (Actual); Last update posted 2022-02-17 (Actual); Status verified 2022-01

CONDITIONS: Infertility, Female
MeSH Terms: conditions — Infertility, Female | interventions — Dydrogesterone; Gonadotropins; Menotropins; Triptorelin Pamoate; Chorionic Gonadotropin; Contraceptives, Oral, Combined; Progesterone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- the progestin primed double stimulation group (Active Comparator): luteal phase priming using combined contraceptive pills from day 21 of the previous cycle for one week by Gynera tab. Controlled ovarian hyper-stimulation with 225-375 IU of gonadotropins will be started day 2-3 of menses after vaginal ultrasound confirming the absence of ovarian cysts. Duphaston at 20 mg/day will be started from the first day of the ovulation induction.Decapeptyl in a dose of 2 ampules of 0.2 mg will be administered when leading follicle >18 mm in diameter for triggering.Then, Controlled ovarian hyper-stimulation the next day after the previous oocyte pickup simultaneously with Duphaston. Starting from the next menstrual cycle Day 3, patients will receive oral estradiol valerate (Cyclo-Progynova (white tablets) daily.When endometrial thickness ≥ 7 mm.Embryo transfer will be scheduled on Day 3, 4 or 5 with maximum number of 3 class A embryos whether of cleavage or blastocyst stage.
  Interventions: Drug: Duphaston; Drug: Gonadotropin; Drug: Decapeptyl; Drug: Combined Oral Contraceptive; Drug: Cyclo-Progynova; Drug: progesterone
- the flexible GnRh antagonist (Active Comparator): This step will be done twice in two different cycles In each cycle: luteal phase priming using combined contraceptive pills from day 21 of the previous cycle for one week by Gynera tab. Controlled ovarian hyper-stimulation using antagonist protocol will be used. Stimulation with 225-375 IU of gonadotropins will be started day 2-3 of menses after vaginal ultrasound confirming the absence of ovarian cysts. Cetrotide ampule will be given daily as the biggest oocyte reaches size 14 mm. Decapeptyl ampules 0.2 mg will be administered when leading follicle >18 mm in diameter. While in the second cycle HCG triggering (Choriomon)in a dose of 10,000 IU will be administered when the leading follicle >18 mm in diameter. Embryo transfer will be scheduled on Day 3, 4 or 5 with maximum number of 3 class A embryos whether of cleavage or blastocyst stage that will be a mixture of the thawed embryos of the first cycle and fresh embryos of the second cycle.
  Interventions: Drug: Gonadotropin; Drug: Cetrotide Injectable Product; Drug: Decapeptyl; Drug: Chorionic Gonadotropin; Drug: Combined Oral Contraceptive; Drug: Cyclo-Progynova; Drug: progesterone

INTERVENTIONS:
Drug: Duphaston — will be used for pituitary suppression in the first arm:20 mg/day will be started from the first day of the ovulation induction in the follicular phase and in the luteal phase will be started the next day after oocyte pickup at 20 mg/day.
  Arms: the progestin primed double stimulation group
Drug: Gonadotropin — will be used for controlled ovarian hyperstimulation in both arms
  Other Names: Fostimon; Menopure; Menogon; Gonapure
Drug: Cetrotide Injectable Product — will used in the second arm for pituitary suppression in the second group daily when the biggest oocyte reaches size 14 mm till ovulation triggering
  Arms: the flexible GnRh antagonist
Drug: Decapeptyl — will be used for ovulation triggering.in the first arm:in a dose of 2 ampules of 0.2 mg will be administered when leading follicle >18 mm in diameter. in the second arm:in a dose of 2 ampules 0.2 mg will be administered when leading follicle >18 mm in diameter in the first cycle only.
Drug: Chorionic Gonadotropin — will be used in the second cycle of the second arm for ovulation triggering in a dose of 10,000 IU when the leading follicle >18 mm in diameter.
  Other Names: choriomon
  Arms: the flexible GnRh antagonist
Drug: Combined Oral Contraceptive — luteal phase priming from day 21 of the cycle before controlled ovarian stimulation for one week .
  Other Names: Gynera
Drug: Cyclo-Progynova — Starting from cycle Day 3 of the intented cycle for thawed embryo transfer, patients will receive the white tablets of Cyclo-Progynova daily. From Day 10 onwards, endometrium growth will be monitored by transvaginal ultrasound.
Drug: progesterone — in the intended cycle of embryo transfer when endometrial thickness ≥ 7 mm. Progesterone administration (as 800 mg/day vaginal suppositories per day and 100 mg ampule IM every other day) will be continued until pregnancy testing 18 days after embryo transfer and in pregnant cases will continued till the 12 weeks of gestation.
  Other Names: prontogest

SUMMARY:
The worldwide prevalence of primary and secondary infertility is estimated at ~2% and 10.5%, respectively, among women aged 20-44 years and attempting to conceive. Poor ovarian responders (PORs) involve 9-24% of patients undergoing in-vitro fertilization (IVF). proper tailoring of the ovarian stimulation protocol in order to maximize the number of oocytes collected represents a crucial step for them to eventually conceive.

Recent evidence indicates that in the same menstrual cycle, there are multiple follicular recruitment waves. This coincides with the theory that folliculogenesis occurs in a wave-like fashion. Thus, within a single menstrual cycle, there can theoretically be multiple opportunities for a clinician to collect oocytes, as opposed to the conventional single cohort of antral follicles during the follicular phase.

Utilizing this concept, clinicians have been attempting to retrieve oocytes from poor responders using both the follicular-phase stimulation (FPS) and the luteal-phase stimulation (LPS) protocols to increase the number of oocytes collected shorter within shorter period of time. By increasing the number of the retrieved oocytes collected, a better clinical can be assured since there is a clear relationship between the number of oocytes collected and live birth rates across all female age groups.

which protocol is the most effective remains controversial and the efficacy of PPOS in POR compared with that of conventional protocols is unclear.

DETAILED DESCRIPTION:
The study will be conducted on 90 infertile women indicated for ICSI with criteria of poor ovarian response defined by Bologna criteria All participants will be informed about the nature of the study and informed consent will be taken from all of them.

Group 1:45 patients will be given the progestin primed double stimulation protocol.

Group 2: 45 patients will be given the flexible GnRh antagonist follicular controlled ovarian stimulations will be done in 2 cycles.

Written informed consents will be obtained from all participants who accept to participate in the research protocol.

Work up:

1. Complete history taking and full assessment of different infertility factors.
2. Hormonal investigations

   * FSH, LH, E2, Prolactin
   * AMH, TSH
3. Basal transvaginal ultrasound

Clinical and embryological procedures:

Group 1:

I. The follicular phase of the double stimulation protocol

1. luteal phase priming using combined contraceptive pills from day 21 of the previous cycle for one week (0.03 mg ethinyl estradiol, gestodene 0.075 mg, Gynera tab, Bayer Pharma AG., Berlin, Germany).
2. Controlled ovarian hyper-stimulation with 225-375 IU of gonadotropins will be started day 2-3 of menses after vaginal ultrasound confirming the absence of ovarian cysts.
3. Dydrogesterone (Duphaston, Abbott company, Illinois, United states) at 20 mg/day will be started from the first day of the ovulation induction.
4. Patient response will be monitored by:

   1. Transvaginal follicular scanning and the dose of the gonadotropins will be modified according to the response.
   2. Serum estradiol.
   3. Serum progesterone and LH on the day of triggering.
5. GnRh agonist triggering (Decapeptyl, Ferring, SAINT-PREX Switzerland) in a dose of 2 ampules of 0.2 mg will be administered when leading follicle >18 mm in diameter.
6. Oocyte pickup will be done 36 hours after GnRh administration with precaution of leaving the follicles measuring 11 mm or less.
7. After the pick-up, oocytes will be denuded. The denuded oocytes are then assessed for nuclear status. Mature oocytes will be used for ICSI.

II. The luteal phase of the double stimulation protocol

Controlled ovarian hyper-stimulation with 225-375 IU of gonadotropins will be started the next day after the previous oocyte pickup simultaneously with Dydrogesterone (Duphaston, Abbott company, Illinois, United states) at 20 mg/day.

The rest will be as the follicular phase.

III. Fertilization and embryo quality:

The fertilization check, which will be performed 16 to 20 hours after ICSI. The resultant embryos will be scored, and they will be vitrified for subsequent transfer.

IV. Embryo transfer

- Starting from the next menstrual cycle Day 3, patients will receive oral estradiol valerate (Cyclo-Progynova (white tablets); Bayer, Germany) daily. From Day 10 onwards, endometrium growth will be monitored by transvaginal ultrasound. When endometrial thickness ≥ 7 mm. Progesterone administration (as 800 mg/day vaginal suppositories per day and 100 mg ampule IM every other day) will be initiated and Embryo transfer will be scheduled on Day 3, 4 or 5 with maximum number of 3 class A embryos whether of cleavage or blastocyst stage.

V. Luteal support - Progesterone administration (as 800 mg/day vaginal suppositories per day and 100 mg ampule IM every other day) will be continued until pregnancy testing 18 days after embryo transfer. The pregnant cases will continue the luteal support till the 12 weeks of gestation.

Group 2:

VI. The flexible GnRH antagonist protocol controlled ovarian stimulation This controlled ovarian stimulation will be done twice in two different cycles

In each cycle:

1. luteal phase priming using combined contraceptive pills from day 21 of the previous cycle for one week (0.03 mg ethinyl estradiol, gestodene 0.075 mg , Gynera tab, Bayer Pharma AG., Berlin, Germany).
2. Controlled ovarian hyper-stimulation using antagonist protocol will be used. Stimulation with 225-375 IU of gonadotropins will be started day 2-3 of menses after vaginal ultrasound confirming the absence of ovarian cysts.
3. GnRH antagonist ( Cetrotide , Merck Serono, Darmstadt, Germany) will be given daily as the biggest oocyte reaches size 14 mm.
4. Patient response will be monitored by:

   1. Transvaginal follicular scanning and the dose of the gonadotropins will be modified according to the response.
   2. Serum estradiol.
   3. Serum progesterone on the day of triggering.
5. GnRh agonist triggering (Decapeptyl, Ferring, Saint-Prex Switzerland) in a dose of 2 ampules 0.2 mg will be administered when leading follicle >18 mm in diameter. While in the second cycle HCG triggering (Choriomon, IBSA, Lugano, Switzerland) in a dose of 10,000 IU will be administered when the leading follicle >18 mm in diameter.
6. Oocyte pickup will be done 36 hours after GnRh administration.
7. After the pick-up, oocytes will be denuded. The denuded oocytes are then assessed for nuclear status. Mature oocytes will be used for ICSI.

VII. Fertilization and embryo quality:

The fertilization check, which will be performed 16 to 20 hours after ICSI. The resultant embryos will be scored.

Embryos of the first cycle will be vitrified while embryos of the second cycle will be freshly transferred unless there is excess for vitrification for subsequent trials of transfer.

VIII. Embryo transfer

- Progesterone administration (as 800 mg/day vaginal suppositories per day and 100 mg ampule IM every other day) will be initiated on the day of the oocyte pick up of the second cycle. Embryo transfer will be scheduled on Day 3, 4 or 5 with maximum number of 3 class A embryos whether of cleavage or blastocyst stage that will be a mixture of the thawed embryos of the first cycle and fresh embryos of the second cycle.

IX. Luteal support Progesterone administration (as 800 mg/day vaginal suppositories per day and 100 mg ampule IM every other day) will be continued until pregnancy testing 18 days after embryo transfer. The pregnant cases will continue the luteal support till the 12 weeks of gestation.

ELIGIBILITY:
Inclusion Criteria:

poor ovarian responders patients defined by Bologna criteria

Exclusion Criteria:

1. Male factor infertility due to azoospermia.
2. Patients with uncorrected uterine pathology.
3. Patients with the diagnosis of severe endometriosis.
4. Patients with BMI over 35.

Ages: 20 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 90 (Actual)
Dates: Start 2020-09-01 (Actual); Primary Completion 2021-03-01 (Actual); Study Completion 2021-09-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Aly A Hussein, Ass.lecturer, Principal Investigator — Elshatby University hospital; Sherif S Gaafar, Professor, Principal Investigator — Elshatby University hospital
Locations (1):
- Elshatby University Maternity Hospital, Alexandria, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Mascarenhas MN, Flaxman SR, Boerma T, Vanderpoel S, Stevens GA. National, regional, and global trends in infertility prevalence since 1990: a systematic analysis of 277 health surveys. PLoS Med. 2012;9(12):e1001356. doi: 10.1371/journal.pmed.1001356. Epub 2012 Dec 18. PMID 23271957
- [Background] Briggs R, Kovacs G, MacLachlan V, Motteram C, Baker HW. Can you ever collect too many oocytes? Hum Reprod. 2015 Jan;30(1):81-7. doi: 10.1093/humrep/deu272. Epub 2014 Oct 31. PMID 25362088
- [Background] Drakopoulos P, Blockeel C, Stoop D, Camus M, de Vos M, Tournaye H, Polyzos NP. Conventional ovarian stimulation and single embryo transfer for IVF/ICSI. How many oocytes do we need to maximize cumulative live birth rates after utilization of all fresh and frozen embryos? Hum Reprod. 2016 Feb;31(2):370-6. doi: 10.1093/humrep/dev316. Epub 2016 Jan 2. PMID 26724797
- [Background] Baerwald AR, Adams GP, Pierson RA. Ovarian antral folliculogenesis during the human menstrual cycle: a review. Hum Reprod Update. 2012 Jan-Feb;18(1):73-91. doi: 10.1093/humupd/dmr039. Epub 2011 Nov 8. PMID 22068695
- [Background] Vanden Brink H, Chizen D, Hale G, Baerwald A. Age-related changes in major ovarian follicular wave dynamics during the human menstrual cycle. Menopause. 2013 Dec;20(12):1243-54. doi: 10.1097/GME.0b013e31828cfb62. PMID 23571519
- [Background] Kuang Y, Chen Q, Hong Q, Lyu Q, Ai A, Fu Y, Shoham Z. Double stimulations during the follicular and luteal phases of poor responders in IVF/ICSI programmes (Shanghai protocol). Reprod Biomed Online. 2014 Dec;29(6):684-91. doi: 10.1016/j.rbmo.2014.08.009. Epub 2014 Sep 6. PMID 25444501
- [Background] Zhang J. Luteal phase ovarian stimulation following oocyte retrieval: is it helpful for poor responders? Reprod Biol Endocrinol. 2015 Jul 25;13:76. doi: 10.1186/s12958-015-0076-2. PMID 26209449
- [Background] Liu C, Jiang H, Zhang W, Yin H. Double ovarian stimulation during the follicular and luteal phase in women >/=38 years: a retrospective case-control study. Reprod Biomed Online. 2017 Dec;35(6):678-684. doi: 10.1016/j.rbmo.2017.08.019. Epub 2017 Aug 24. PMID 29030068
- [Background] Zhang Q, Guo XM, Li Y. Implantation rates subsequent to the transfer of embryos produced at different phases during double stimulation of poor ovarian responders. Reprod Fertil Dev. 2017 Jun;29(6):1178-1183. doi: 10.1071/RD16020. PMID 27166216
- [Background] Sunkara SK, Rittenberg V, Raine-Fenning N, Bhattacharya S, Zamora J, Coomarasamy A. Association between the number of eggs and live birth in IVF treatment: an analysis of 400 135 treatment cycles. Hum Reprod. 2011 Jul;26(7):1768-74. doi: 10.1093/humrep/der106. Epub 2011 May 10. PMID 21558332
- [Background] Wang N, Wang Y, Chen Q, Dong J, Tian H, Fu Y, Ai A, Lyu Q, Kuang Y. Luteal-phase ovarian stimulation vs conventional ovarian stimulation in patients with normal ovarian reserve treated for IVF: a large retrospective cohort study. Clin Endocrinol (Oxf). 2016 May;84(5):720-8. doi: 10.1111/cen.12983. Epub 2015 Dec 21. PMID 26603821
- [Background] McNatty KP, Hillier SG, van den Boogaard AM, Trimbos-Kemper TC, Reichert LE Jr, van Hall EV. Follicular development during the luteal phase of the human menstrual cycle. J Clin Endocrinol Metab. 1983 May;56(5):1022-31. doi: 10.1210/jcem-56-5-1022. PMID 6403567
- [Background] Moffat R, Pirtea P, Gayet V, Wolf JP, Chapron C, de Ziegler D. Dual ovarian stimulation is a new viable option for enhancing the oocyte yield when the time for assisted reproductive technnology is limited. Reprod Biomed Online. 2014 Dec;29(6):659-61. doi: 10.1016/j.rbmo.2014.08.010. Epub 2014 Sep 4. PMID 25311972
- [Background] Kuang Y, Chen Q, Fu Y, Wang Y, Hong Q, Lyu Q, Ai A, Shoham Z. Medroxyprogesterone acetate is an effective oral alternative for preventing premature luteinizing hormone surges in women undergoing controlled ovarian hyperstimulation for in vitro fertilization. Fertil Steril. 2015 Jul;104(1):62-70.e3. doi: 10.1016/j.fertnstert.2015.03.022. Epub 2015 May 5. PMID 25956370
- [Background] Ferraretti AP, La Marca A, Fauser BC, Tarlatzis B, Nargund G, Gianaroli L; ESHRE working group on Poor Ovarian Response Definition. ESHRE consensus on the definition of 'poor response' to ovarian stimulation for in vitro fertilization: the Bologna criteria. Hum Reprod. 2011 Jul;26(7):1616-24. doi: 10.1093/humrep/der092. Epub 2011 Apr 19. PMID 21505041

RESULTS

PARTICIPANT FLOW:
Groups:
- the Progestin Primed Double Stimulation Group: luteal phase priming using combined contraceptive pills from day 21 of the previous cycle for one week by Gynera tab. Controlled ovarian hyper-stimulation with 225-375 IU of gonadotropins will be started day 2-3 of menses after vaginal ultrasound confirming the absence of ovarian cysts. Duphaston at 20 mg/day will be started from the first day of the ovulation induction.Decapeptyl in a dose of 2 ampules of 0.2 mg will be administered when leading follicle >18 mm in diameter for triggering.Oocyte pickup will be done 36 hours after GnRh administration . The resultant embryos will be scored, and they will be vitrified for subsequent transfer.Then, Controlled ovarian hyper-stimulation the next day after the previous oocyte pickup simultaneously with Duphaston. .Decapeptyl in a dose of 2 ampules of 0.2 mg will be administered when leading follicle >18 mm in diameter for triggering.Oocyte pickup will be done 36 hours after GnRh administration The resultant embryos will be scored, and they will be vitrified for subsequent transfer.Starting from the next menstrual cycle Day 3, patients will receive oral estradiol valerate (Cyclo-Progynova (white tablets) daily.When endometrial thickness ≥ 7 mm.Embryo transfer will be scheduled on Day 3, 4 or 5 with maximum number of 3 class A embryos whether of cleavage or blastocyst stage.
- the Flexible GnRh Antagonist: This step will be done twice in two different cycles In each cycle: luteal phase priming using combined contraceptive pills from day 21 of the previous cycle for one week by Gynera tab. Controlled ovarian hyper-stimulation using antagonist protocol will be used. Stimulation with 225-375 IU of gonadotropins will be started day 2-3 of menses after vaginal ultrasound confirming the absence of ovarian cysts. Cetrotide ampule will be given daily as the biggest oocyte reaches size 14 mm. Decapeptyl ampules 0.2 mg will be administered when leading follicle >18 mm in diameter.Oocyte pickup will be done 36 hours after GnRh administration. Embryos of the first cycle will be vitrified . . While in the second cycle HCG triggering (Choriomon)in a dose of 10,000 IU will be administered when the leading follicle >18 mm in diameter. Oocyte pickup will be done 36 hours after GnRh administration . embryos of the second cycle will be freshly transferred unless there is excess so being verified for subsequent transfer.Starting from the next menstrual cycle Day 3, patients will receive oral estradiol valerate (Cyclo-Progynova (white tablets) daily.When endometrial thickness ≥ 7 mm.Embryo transfer will be scheduled on Day 3, 4 or 5 with maximum number of 3 class A embryos whether of cleavage or blastocyst stage that will be a mixture of the thawed embryos of the first cycle and fresh embryos of the second cycle.
  .
Period: Overall Study
Arm/Group | the Progestin Primed Double Stimulation Group | the Flexible GnRh Antagonist
Started | 45 | 45
Completed | 41 | 42
Not Completed | 4 | 3
Not completed — Protocol Violation | 3 | 2
Not completed — Lost to Follow-up | 1 | 0
Not completed — Withdrawal by Subject | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | the Progestin Primed Double Stimulation Group | the Flexible GnRh Antagonist | Total
Number analyzed (Participants) | 41 | 42 | 83
Age, Continuous [Mean (Standard Deviation); unit: years] | 34.05 (5) | 35.48 (6.99) | 34.77 (6.09)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 41 | 42 | 83
  Male | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 41 | 42 | 83
Region of Enrollment [Number; unit: participants]
  Egypt | 41 | 42 | 83
duration of infertility [Median (Inter-Quartile Range); unit: years] | 5 [3 to 6] | 5 [2 to 8] | 5 [2 to 7]
previous ICSI trials [Number; unit: participants]
  had no previous ICSI trials | 22 | 26 | 48
  had 1 failed ICSI trial | 17 | 14 | 31
  had 2 failed ICSI trials | 2 | 2 | 4

OUTCOME MEASURES:

1. Primary Outcome: the Number of M2 Oocytes Retrieved
Description: it is the number of M2 oocytes retrieved that were being assessed after denudation
Time Frame: 1-2 hours after oocyte retrieval
Measure: Median (Inter-Quartile Range); unit: oocytes
Groups:
- the Progestin Primed Double Stimulation Group: luteal phase priming using combined contraceptive pills from day 21 of the previous cycle for one week by Gynera tab. Controlled ovarian hyper-stimulation with 225-375 IU of gonadotropins will be started day 2-3 of menses after vaginal ultrasound confirming the absence of ovarian cysts. Duphaston 20 mg/day will be started from the first day of the ovulation induction.Decapeptyl in a dose of 2 ampules of 0.2 mg will be administered when leading follicle >18 mm in diameter for triggering.Oocyte pickup will be done 36 hours after GnRh administration . The resultant embryos will be scored, and they will be vitrified for subsequent transfer.Then, Controlled ovarian hyper-stimulation the next day after the previous oocyte pickup simultaneously with Duphaston. .Decapeptyl in a dose of 2 ampules of 0.2 mg will be administered when leading follicle >18 mm in diameter for triggering.Oocyte pickup will be done 36 hours after GnRh administration The resultant embryos will be scored, and they will be vitrified for subsequent transfer.Starting from the next menstrual cycle Day 3, patients will receive oral estradiol valerate (Cyclo-Progynova (white tablets) daily.When endometrial thickness ≥ 7 mm.Embryo transfer will be scheduled on Day 3, 4 or 5 with maximum number of 3 class A embryos whether of cleavage or blastocyst stage.
- the Flexible GnRh Antagonist Group: This step will be done twice in two different cycles In each cycle: luteal phase priming using combined contraceptive pills from day 21 of the previous cycle for one week by Gynera tab. Controlled ovarian hyper-stimulation using antagonist protocol will be used. Stimulation with 225-375 IU of gonadotropins will be started day 2-3 of menses after vaginal ultrasound confirming the absence of ovarian cysts. Cetrotide ampule will be given daily as the biggest oocyte reaches size 14 mm. Decapeptyl ampules 0.2 mg will be administered when leading follicle >18 mm in diameter.Oocyte pickup will be done 36 hours after GnRh administration. Embryos of the first cycle will be vitrified . While in the second cycle HCG triggering (Choriomon)in a dose of 10,000 IU will be administered when the leading follicle >18 mm in diameter. Oocyte pickup will be done 36 hours after GnRh administration . embryos of the second cycle will be freshly transferred unless there is excess so being verified for subsequent transfer.Starting from the next menstrual cycle Day 3, patients will receive oral estradiol valerate (Cyclo-Progynova (white tablets) daily.When endometrial thickness ≥ 7 mm.Embryo transfer will be scheduled on Day 3, 4 or 5 with maximum number of 3 class A embryos whether of cleavage or blastocyst stage that will be a mixture of the thawed embryos of the first cycle and fresh embryos of the second cycle.
Arm/Group | the Progestin Primed Double Stimulation Group | the Flexible GnRh Antagonist Group
Number analyzed (Participants) | 41 | 42
oocytes | 6 [3 to 7] | 4.5 [3 to 8]
Statistical Analysis 1: Comparison: the Progestin Primed Double Stimulation Group vs the Flexible GnRh Antagonist Group; Test type: Other; p = 0.254, Wilcoxon (Mann-Whitney); Median Difference (Final Values) = 1.5

2. Primary Outcome: the Fertilization Rate
Description: percentage transformation of micro injected oocytes into two pronuclei. it is done 16 to 20 hours after microinjection of the oocytes by the sperms
Time Frame: 16 to 20 hours after microinjection of the oocytes with the sperms
Measure: Median (Inter-Quartile Range); unit: percentage of transformation
Arm/Group | the Progestin Primed Double Stimulation Group | the Flexible GnRh Antagonist Group
Number analyzed (Participants) | 41 | 42
percentage of transformation | 71.43 [66.67 to 100] | 80.91 [66.67 to 100]
Statistical Analysis 1: Comparison: the Progestin Primed Double Stimulation Group vs the Flexible GnRh Antagonist Group; Test type: Other; p = 0.219, Wilcoxon (Mann-Whitney); Median Difference (Final Values) = 9.48

3. Primary Outcome: the Resultant Embryos Number
Description: it is the resultant embryos number counted day 3 or 4 or 5 after fertilization
Time Frame: the embryos number counted day 3 or 4or 5 after fertilization
Measure: Median (Inter-Quartile Range); unit: number of embryos
Arm/Group | the Progestin Primed Double Stimulation Group | the Flexible GnRh Antagonist Group
Number analyzed (Participants) | 41 | 42
number of embryos | 4 [3 to 5] | 3 [2 to 6]
Statistical Analysis 1: Comparison: the Progestin Primed Double Stimulation Group vs the Flexible GnRh Antagonist Group; Test type: Other; p = 0.269, Wilcoxon (Mann-Whitney); Median Difference (Final Values) = 1

4. Primary Outcome: the Implantation Rate
Description: it is calculated as the number of intrauterine gestational sacs observed by transvaginal ultrasonography divided by the number of transferred embryos at the 6 th week of pregnancy and then multiplied by 100
Time Frame: at the 6 th week of pregnancy
Measure: Median (Inter-Quartile Range); unit: percentage
Arm/Group | the Progestin Primed Double Stimulation Group | the Flexible GnRh Antagonist Group
Number analyzed (Participants) | 7 | 8
percentage | 50 [50 to 100] | 50 [33.33 to 50]
Statistical Analysis 1: Comparison: the Progestin Primed Double Stimulation Group vs the Flexible GnRh Antagonist Group; Test type: Other; p = 0.072, Wilcoxon (Mann-Whitney); Median Difference (Final Values) = 0

5. Primary Outcome: the Clinical Pregnancy Rate.
Description: percentage of cases in which observation of a gestational sac with fetal heart beat by transvaginal ultrasound at 6 weeks of pregnancy
Time Frame: at the 6 th weeks of pregnancy
Measure: Number; unit: percentage of participants
Arm/Group | the Progestin Primed Double Stimulation Group | the Flexible GnRh Antagonist Group
Number analyzed (Participants) | 41 | 42
percentage of participants | 7 | 8
Statistical Analysis 1: Comparison: the Progestin Primed Double Stimulation Group vs the Flexible GnRh Antagonist Group; Test type: Other; p = 1, Fisher Exact

6. Secondary Outcome: the Difference in the Ongoing Pregnancy Rate in Both Protocols.
Description: Assessing the difference in the ongoing pregnancy rate when the pregnancy had completed ≥20 weeks of gestation
Time Frame: At the 20 th week of gestation
Measure: Number; unit: percentage of participants
Arm/Group | the Progestin Primed Double Stimulation Group | the Flexible GnRh Antagonist Group
Number analyzed (Participants) | 41 | 42
percentage of participants | 6 | 5
Statistical Analysis 1: Comparison: the Progestin Primed Double Stimulation Group vs the Flexible GnRh Antagonist Group; Test type: Other; p = 0.720, Chi-squared

7. Secondary Outcome: the Difference Between the Follicular Phase and the Luteal Phase of the Progestin Primed Double Stimulation Protocol Regarding the Total Days of Controlled Ovarian Hyperstimulation
Description: the total number of days of the controlled ovarian hyperstimulation in both follicular and luteal phase of the progestin primed double stimulation protocol are studied so as to asses the difference between the two phases, the follicular phase and the luteal phase of the progestin primed double stimulation protocol
Time Frame: From the first day of ovarian stimulation till the last day of ovarian stimulation in each phase ,the follicular and the luteal, of stimulation
Population: the progestin primed dual stimulation group are subdivided into the follicular phase stimulation and the luteal phase stimulation so as to study the difference between both phases
Measure: Median (Inter-Quartile Range); unit: number of days
Groups:
- the Follicular Phase of the Progestin Primed Double Stimulation Group: luteal phase priming using combined contraceptive pills from day 21 of the previous cycle for one week by Gynera tab. Controlled ovarian hyper-stimulation with 225-375 IU of gonadotropins will be started day 2-3 of menses after vaginal ultrasound confirming the absence of ovarian cysts. Duphaston at 20 mg/day will be started from the first day of the ovulation induction.Decapeptyl in a dose of 2 ampules of 0.2 mg will be administered when leading follicle >18 mm in diameter for triggering.Oocyte pickup will be done 36 hours after GnRh administration. The resultant embryos will be scored, and they will be vitrified for subsequent transfer
- the Luteal Phase of the Progestin Primed Double Stimulation Group: Controlled ovarian hyper-stimulation the next day after the previous oocyte pickup simultaneously with Duphaston. .Decapeptyl in a dose of 2 ampules of 0.2 mg will be administered when leading follicle >18 mm in diameter for triggering.Oocyte pickup will be done 36 hours after GnRh administration The resultant embryos will be scored, and they will be vitrified for subsequent transfer
Arm/Group | the Follicular Phase of the Progestin Primed Double Stimulation Group | the Luteal Phase of the Progestin Primed Double Stimulation Group
Number analyzed (Participants) | 41 | 41
number of days | 10 [9 to 12] | 12 [10 to 13]
Statistical Analysis 1: Comparison: the Follicular Phase of the Progestin Primed Double Stimulation Group vs the Luteal Phase of the Progestin Primed Double Stimulation Group; Test type: Other; p = 0.002, Wilcoxon (Mann-Whitney); Median Difference (Final Values) = 2

8. Secondary Outcome: the Difference Between the Follicular Phase and the Luteal Phase of the Progestin Primed Double Stimulation Protocol Regarding the Total Dosage of Gonadotropins Used in the Controlled Ovarian Hyperstimulation
Description: Assessing the difference between the follicular phase and the luteal phase of the progestin primed double stimulation protocol regarding the total dosage of gonadotropins used in the controlled ovarian hyperstimulation so as to the difference between the two phases
Time Frame: as for outcome 7
Population: as for outcome 7
Measure: Median (Inter-Quartile Range); unit: IU
Arm/Group | the Follicular Phase of the Progestin Primed Double Stimulation Group | the Luteal Phase of the Progestin Primed Double Stimulation Group
Number analyzed (Participants) | 41 | 41
IU | 3000 [2700 to 3150] | 3600 [3000 to 3750]
Statistical Analysis 1: Comparison: the Follicular Phase of the Progestin Primed Double Stimulation Group vs the Luteal Phase of the Progestin Primed Double Stimulation Group; Test type: Other; p = 0.007, Wilcoxon (Mann-Whitney); Median Difference (Final Values) = 600

9. Secondary Outcome: the Difference Between the Follicular Phase and the Luteal Phase of the Progestin Primed Double Stimulation Protocol Regarding the Number of M2 Oocytes Retrieved
Description: it is the number of M2 oocytes retrieved that were being assessed after denudation so as to the difference between the results between the two phases, the follicular phase and the luteal phase of the progestin primed double stimulation protocol
Time Frame: 1-2 hours after oocyte retrieval
Population: as for outcome 7
Measure: Median (Inter-Quartile Range); unit: number of oocytes
Arm/Group | the Follicular Phase of the Progestin Primed Double Stimulation Group | the Luteal Phase of the Progestin Primed Double Stimulation Group
Number analyzed (Participants) | 41 | 41
number of oocytes | 2 [1 to 3] | 4 [2 to 5]
Statistical Analysis 1: Comparison: the Follicular Phase of the Progestin Primed Double Stimulation Group vs the Luteal Phase of the Progestin Primed Double Stimulation Group; Test type: Other; p = 0.001, Wilcoxon (Mann-Whitney); Median Difference (Final Values) = 2

10. Secondary Outcome: the Difference Between the Follicular Phase and the Luteal Phase of the Progestin Primed Double Stimulation Protocol Regarding the Fertilization Rate.
Description: percentage of transformation of micro injected oocytes into two pronuclei at 16 -20 hours after microinjection of the oocytes by the sperms so as to the difference between the results between the two phases, the follicular phase and the luteal phase of the progestin primed double stimulation protocol
Time Frame: 16 to 20 hours after microinjection of the oocytes with the sperms
Population: as for outcome 7
Measure: Median (Inter-Quartile Range); unit: percentage
Groups:
- the Follicular Phase of the Progestin Primed Double Stimulation Group: luteal phase priming using combined contraceptive pills from day 21 of the previous cycle for one week by Gynera tab. Controlled ovarian hyper-stimulation with 225-375 IU of gonadotropins will be started day 2-3 of menses after vaginal ultrasound confirming the absence of ovarian cysts. Duphaston at 20 mg/day will be started from the first day of the ovulation induction.Decapeptyl in a dose of 2 ampules of 0.2 mg will be administered when leading follicle >18 mm in diameter for triggering.Oocyte pickup will be done 36 hours after GnRh administration . The resultant embryos will be scored, and they will be vitrified for subsequent transfer
- the Luteal Phase of the Progestin Primed Double Stimulation Group: Controlled ovarian hyper-stimulation the next day after the previous oocyte pickup simultaneously with Duphaston.Decapeptyl in a dose of 2 ampules of 0.2 mg will be administered when leading follicle >18 mm in diameter for triggering.Oocyte pickup will be done 36 hours after GnRh administration The resultant embryos will be scored, and they will be vitrified for subsequent transfer
Arm/Group | the Follicular Phase of the Progestin Primed Double Stimulation Group | the Luteal Phase of the Progestin Primed Double Stimulation Group
Number analyzed (Participants) | 41 | 41
percentage | 66.67 [50 to 100] | 100 [60 to 100]
Statistical Analysis 1: Comparison: the Follicular Phase of the Progestin Primed Double Stimulation Group vs the Luteal Phase of the Progestin Primed Double Stimulation Group; Test type: Other; p = 0.04, Wilcoxon (Mann-Whitney); Median Difference (Final Values) = 33.33

11. Secondary Outcome: the Difference Between the Follicular Phase and the Luteal Phase of the Progestin Primed Double Stimulation Protocol Regarding the Resultant Embryos Number
Description: the resultant embryos number are counted day 3 or 4 or 5 after fertilization so as to the difference between the results between the two phases, the follicular phase and the luteal phase of the progestin primed double stimulation protocol
Time Frame: the embryos number counted day 3 or 4or 5 after fertilization
Population: as for outcome 7
Measure: Median (Inter-Quartile Range); unit: number of embryos
Arm/Group | the Follicular Phase of the Progestin Primed Double Stimulation Group | the Luteal Phase of the Progestin Primed Double Stimulation Group
Number analyzed (Participants) | 41 | 42
number of embryos | 1 [1 to 2] | 3 [2 to 4]
Statistical Analysis 1: Comparison: the Follicular Phase of the Progestin Primed Double Stimulation Group vs the Luteal Phase of the Progestin Primed Double Stimulation Group; Test type: Other; p < 0.001, Wilcoxon (Mann-Whitney); Median Difference (Final Values) = 2

12. Secondary Outcome: Assessing the Difference Between the Follicular Phase of the Progestin Primed Double Stimulation Protocol and the First Round of the Conventional GnRH Antagonist Protocol Regarding the Number of M2 Oocytes Retrieved .
Description: it is the number of M2 oocytes retrieved that were being assessed after denudation.so as to study the effect of the progestin used on the ovarian response in poor ovarian responders, we have compared the follicular phase of the dual stimulation group and first follicular wave of the flexible antagonist group
Time Frame: 1-2 hours after oocyte retrieval
Population: as for outcome 7
Measure: Median (Inter-Quartile Range); unit: number of oocytes
Groups:
- The Follicular Phase of the Double Stimulation Group: luteal phase priming using combined contraceptive pills from day 21 of the previous cycle for one week by Gynera tab. Controlled ovarian hyper-stimulation with 225-375 IU of gonadotropins will be started day 2-3 of menses after vaginal ultrasound confirming the absence of ovarian cysts. Duphaston at 20 mg/day will be started from the first day of the ovulation induction.Decapeptyl in a dose of 2 ampules of 0.2 mg will be administered when leading follicle >18 mm in diameter for triggering.Oocyte pickup will be done 36 hours after GnRh administration . The resultant embryos will be scored, and they will be vitrified for subsequent transfer
- the First Round of the Conventional GnRH Antagonist Group: luteal phase priming using combined contraceptive pills from day 21 of the previous cycle for one week by Gynera tab. Controlled ovarian hyper-stimulation using antagonist protocol will be used. Stimulation with 225-375 IU of gonadotropins will be started day 2-3 of menses after vaginal ultrasound confirming the absence of ovarian cysts. Cetrotide ampule will be given daily as the biggest oocyte reaches size 14 mm. Decapeptyl ampules 0.2 mg will be administered when leading follicle >18 mm in diameter.Oocyte pickup will be done 36 hours after GnRh administration. Embryos of the first cycle will be vitrified
Arm/Group | The Follicular Phase of the Double Stimulation Group | the First Round of the Conventional GnRH Antagonist Group
Number analyzed (Participants) | 41 | 42
number of oocytes | 2 [1 to 3] | 2 [1 to 3]
Statistical Analysis 1: Comparison: The Follicular Phase of the Double Stimulation Group vs the First Round of the Conventional GnRH Antagonist Group; Test type: Other; p = 0.851, Wilcoxon (Mann-Whitney); Median Difference (Final Values) = 0

13. Secondary Outcome: Assessing the Difference Between the Follicular Phase of the Progestin Primed Double Stimulation Protocol and the First Round of the Conventional GnRH Antagonist Protocol Regarding the Fertilization Rate.
Description: it is percentage transformation of micro injected oocytes into two pronuclei.so as to study the effect of the progestin used on the ovarian response and its results in poor ovarian responders, we have compared the follicular phase of the dual stimulation group and first follicular wave of the flexible antagonist group
Time Frame: 16 to 20 hours after microinjection of the oocytes by the sperms
Measure: Median (Inter-Quartile Range); unit: percentage
Arm/Group | The Follicular Phase of the Double Stimulation Group | the First Round of the Conventional GnRH Antagonist Group
Number analyzed (Participants) | 41 | 42
percentage | 66.67 [50 to 100] | 91.67 [50 to 100]
Statistical Analysis 1: Comparison: The Follicular Phase of the Double Stimulation Group vs the First Round of the Conventional GnRH Antagonist Group; Test type: Other; p = 0.304, Wilcoxon (Mann-Whitney); Median Difference (Final Values) = 25

14. Secondary Outcome: Assessing the Difference Between the Follicular Phase of the Progestin Primed Double Stimulation Protocol and the First Round of the Conventional GnRH Antagonist Protocol Regarding the Resultant Embryos Number.
Description: it is the number of the resultant embryos counted at day 3 or 4 or 5 after fertilization.so as to study the effect of the progestin used on the ovarian response and the resultant embryos number in poor ovarian responders, we have compared the follicular phase of the dual stimulation group and first follicular wave of the flexible antagonist group
Time Frame: at day 3 or 4or 5 after fertilization
Measure: Mean (Standard Deviation); unit: percentage
Arm/Group | The Follicular Phase of the Double Stimulation Group | the First Round of the Conventional GnRH Antagonist Group
Number analyzed (Participants) | 41 | 42
percentage | 1.66 (1.44) | 1.69 (1.18)
Statistical Analysis 1: Comparison: The Follicular Phase of the Double Stimulation Group vs the First Round of the Conventional GnRH Antagonist Group; Test type: Other; p = 0.486, Wilcoxon (Mann-Whitney); Median Difference (Final Values) = 1

ADVERSE EVENTS:
Time Frame: from the 1 st day of ovarian priming prior to ovarian stimulation till the 20th week of pregnancy.
Groups:
- the Progestin Primed Double Stimulation Group: luteal phase priming using combined contraceptive pills from day 21 of the previous cycle for one week by Gynera tab. Controlled ovarian hyper-stimulation with 225-375 IU of gonadotropins will be started day 2-3 of menses after vaginal ultrasound confirming the absence of ovarian cysts. Duphaston at 20 mg/day will be started from the first day of the ovulation induction.Decapeptyl in a dose of 2 ampules of 0.2 mg will be administered when leading follicle >18 mm in diameter for triggering .Then, Controlled ovarian hyper-stimulation the next day after the previous oocyte pickup simultaneously with Duphaston. Starting from the next menstrual cycle Day 3, patients will receive oral estradiol valerate (Cyclo-Progynova (white tablets) daily.When endometrial thickness ≥ 7 mm.Embryo transfer will be scheduled on Day 3, 4 or 5 with maximum number of 3 class A embryos whether of cleavage or blastocyst stage.
Arm/Group | the Progestin Primed Double Stimulation Group | the Flexible GnRh Antagonist
All-Cause Mortality (participants affected / at risk) | 0/41 | 0/42
Serious Adverse Events (participants affected / at risk) | 0/41 | 0/42
Other Adverse Events (participants affected / at risk) | 12/41 | 10/42
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | the Progestin Primed Double Stimulation Group (N=41) | the Flexible GnRh Antagonist (N=42)
nausea and abdominal distention (Gastrointestinal disorders) | 5 (15) | 5 (12)
pelvic pain (Reproductive system and breast disorders) | 3 (10) | 3 (8)
headache (Nervous system disorders) | 4 (10) | 2 (5)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-01-26): https://cdn.clinicaltrials.gov/large-docs/78/NCT04537078/Prot_SAP_001.pdf